CLINICAL TRIAL: NCT00491881
Title: Effect of "no Added Salt Diet " on Blood Pressure Control & 24 Hour Urinary Sodium Excretion in Mild to Moderate Hypertension
Brief Title: Effect of no Added Salt Diet on Urinary Sodium and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2384
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-06

CONDITIONS: Hypertension
Keywords: blood pressure; No added salt diet; urinary sodium
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: no added salt diet

SUMMARY:
There is much evidence that a reduction in dietary salt intake lowers blood pressure in hypertensive individuals, however few have looked at effect of 'no added salt diet' and modest salt intake on total restriction of sodium intake with especial attention to very exact surrogate of urinary sodium excretion. Our study demonstrates that a modest reduction in salt intake from regular level of 10 - 12 g per day to the recommended level of 5 - 6 g per day lowers blood pressure by 12.1/ 6.8 mmHg at day time and 11.1/5.9 mmhg at night time.However only 35% of patients reach to the goal of sodium restriction of diet(below 100 meq/dl in 24 hours urine.It means even modest salt restriction can dramatically decrease blood pressure with no added salt diet.

DETAILED DESCRIPTION:
Abstract Incidence of Hypertension as a major cardiovascular treat is increasing. The best known diet for hypertensives is 'no added salt diet'.

In this study we evaluated the effect of 'no added salt diet' on hypertensive population with high dietary sodium intake by measuring 24 hour urinary sodium excretion.

Method & results: In this single center randomized study 80 patients (60 cases and 20 controls) not on any drug therapy for hypertension with mild to moderate hypertension were enrolled. 24 hour holter monitoring of BP and 24 hour urinary sodium excretion were measured before and after 6 weeks of 'no added salt diet'. There is no statistically significant difference between age , weight , sex , Hyperlipidemia , family history of hypertension , mean systolic & diastolic BP at day and night and mean urinary sodium excretion in 24 hour urine of case &control groups .78% of all patients had moderate to high salt intake .

After 6 week of 'no added salt diet' systolic & diastolic BP significantly decreased at day (mean decrease: 12.1 /6.8 mmhg) and night (mean decrease: 11.1/5.9 mmhg ) which is statistically significant between case & control groups (P 0.0001).

Urinary sodium excretion of 24 hour urine decreased 37.1meq/d ± 39,67mg/dl which is statistically significant in case & control groups (p: 0.0001).

Only 36% of patients after no added salt diet reach to pretreatment goal of 24 hour urinary sodium excretion of below 100meq/dl (P:0.001).

Conclusion: despite modest effect on dietary sodium restriction, no added salt diet significantly decreases systolic & diastolic BP and should be advised to every hypertensive patients. Trial registration research deputy-smums84-2384 Key words: blood pressure, No added salt diet, urinary sodium

ELIGIBILITY:
Inclusion Criteria:

* Hypertension proved by 24 hours holter monitoring
* Mild to moderate hypertension
* Signing the written consent

Exclusion Criteria:

* Use of any drug for hypertension
* Use of any drug for 6 week period
* Unable to collect 24 hours urine
* Unable to tolerate 24 hours holter of blood pressure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2005 (Actual)
Dates: Start 2005-05; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
decrease blood pressure | after 6 weeks of diet

SECONDARY OUTCOMES:
decrease 24 hours urinary sodium excretion | after 6 weeks of diet

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, M.D., Study Director — Shiraz University of Medical Sciences
Locations (1):
- Motahhari outpatient clinic, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kojuri J, Rahimi R. Effect of "no added salt diet" on blood pressure control and 24 hour urinary sodium excretion in mild to moderate hypertension. BMC Cardiovasc Disord. 2007 Nov 6;7:34. doi: 10.1186/1471-2261-7-34. PMID 17986327